CLINICAL TRIAL: NCT04299243
Title: Clinical Trial Protocol for Safety and Efficacy of Soft Contact Lens (Model: Spherical Lens)
Brief Title: Clinical Trial Protocol for Safety and Efficacy of Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLP-01
Record Dates: First submitted 2020-02-18; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spherical Lens (Experimental): Randomized to Spherical Lens worn in a daily disposable mode
  Interventions: Device: Contact Lenses
- SiHy Daily (Active Comparator): Randomized to SiHy Daily worn in a daily disposable mode
  Interventions: Device: Contact Lenses

INTERVENTIONS:
Device: Contact Lenses — Contact lenses for vision correction

SUMMARY:
This project is a multi-center, randomized, parallel-controlled, non-inferior clinical trial of soft contact lenses.

DETAILED DESCRIPTION:
The test product is the Soft Contact Lens (model: Spherical Lens), and the control product is a commercially available soft contact lens (model: SiHy Daily). The number of enrolled subjects is 148, and clinical observation is performed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age of 18 to 45
* Spherical power: -0.25 to -10.00D
* Cylinder power ≤0.75D and Sph.P:Cyl.P≥3:1, or 1.00D≤ cylinder power ≤1.50D and Sph.P:Cyl.P ≥4:1;
* Both eyes are ametropia, and there is no case where the investigator believes that the soft contact lens cannot be worn;

  : The case of wearing a soft contact lens as referred to in this trial is: i) No eyelid abnormalities or infections; ii) No clinically significant slit lamp findings iii) No other active eye diseases.
* BCVA of the left and right eye subjective refraction is greater than or equal to 5.0.

Exclusion Criteria:

* Need to use therapeutic ophthalmic drugs, including antibiotics, hormones and compound ophthalmic drugs containing hormones
* Dry eye syndrome
* Any systemic disease contraindications to contact lenses or disease medications can affect the wearing of contact lenses
* Wearing a hard contact lens in the past 6 weeks
* Tear film break-up time is less than or equal to 5s
* Allergic to contact lenses and/or contact lenses
* Keratoconus or other irregular corneal patients
* Soft hydrophilic contact lens wearers are affected by long-term special conditions such as dryness, severe dust or volatile chemicals
* Pregnant, lactating or plan to be pregnant
* Only one eye meets the requirements for enrollment
* Participating in other clinical trials or less than ten days after the end of a soft contact lens clinical trial
* Less than three months after the end of a drug clinical trial
* Determined by the investigator that could not be enrolled

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The ratio of corrected visual acuity of left and right eyes is ≥5.0 | 1 week
  The standard logarithmic visual acuity chart consistent with the guiding principle is adopted in this scheme.
  - Success criteria: If the lower limit of 95% CI of the evaluated rate of corrected for visual acuity for both eyes ≥ 5.0 at 1 week visit is ≥-10%, the primary endpoint of the two groups is non-inferior.
The occurrence of adverse events | 3 month
  Compare the number of adverse events and serious adverse events, the number of cases and the incidence rate; list the number and cases of adverse events; describe the adverse events that are related to the investigational products.

SECONDARY OUTCOMES:
BCVA (spectacles) and BCVA (CL) | 1 week, 1 month, 3 months
  BCVA (spectacles and CL) of both eyes are compared at baseline and at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Li Lihua, MD, Principal Investigator — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China